CLINICAL TRIAL: NCT03363763
Title: Phase 2 Multi Center Prospective Rand. Double Blind Placebo Cont. Parallel Design Study to Evaluate Safety & Efficacy of Topical Sirolimus for Cutaneous Angiofibromas in Subjects W/ Tuberous Sclerosis Complex Followed by Opt. Open Label
Brief Title: Topical Sirolimus Ointment for Cutaneous Angiofibromas in Subjects With Tuberous Sclerosis Complex
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated (The clinical trial has ended prematurely due to low patient recruitment)
Sponsor: Aucta Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AUCTA-UAP006-PH2
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2025-12-01 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Angiofibroma of Face; Tuberous Sclerosis
Keywords: rash; fibroma; skin; facial; face; bumps; redness; erythema; lesions; papules; blood vessel; cheeks
MeSH Terms: conditions — Tuberous Sclerosis; Exanthema; Fibroma; Facies; Erythema | interventions — Sirolimus

STUDY DESIGN:
Intervention Model Description: Subjects will be randomly assigned in a 1:1:1 ratio to receive 1 of 2 treatments or placebo. The randomization is stratified by site.
  Subjects who complete the double-blind phase of the study with an overall compliance rate >80% and <120%, as determined by weight of returned study medication, will be offered entry into an open-label period for an additional 12 weeks.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Sirolimus 0.2% (Active Comparator): Sirolimus 0.2% ointment applied topically hs x 12 weeks
  Interventions: Drug: Sirolimus 0.2%
- Sirolimus 0.4% (Active Comparator): Sirolimus 0.4% ointment applied topically hs x 12 weeks
  Interventions: Drug: Sirolimus 0.4%
- Placebo (Placebo Comparator): Placebo ointment applied topically hs x 12 weeks
  Interventions: Drug: Placebo ointment

INTERVENTIONS:
Drug: Sirolimus 0.2% — Ointment for topical administration hs x 12 weeks
  Other Names: Rapamune; rapamycin; mTOR inhibitor
  Arms: Sirolimus 0.2%
Drug: Sirolimus 0.4% — Ointment for topical administration hs x 12 weeks
  Other Names: Rapamune; rapamycin; mTOR inhibitor
  Arms: Sirolimus 0.4%
Drug: Placebo ointment — Placebo ointment comparator for topical administration hs x 12 weeks
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of sirolimus (0.2% and 0.4% formulations) and its vehicle when applied topically once daily for 12 weeks for the treatment of cutaneous angiofibromas in pediatric subjects with tuberous sclerosis complex (TSC).

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-blind, placebo-controlled, multicenter study designed to assess the safety and efficacy of topically-applied sirolimus for the treatment of cutaneous angiofibromas in pediatric subjects with TSC. Approximately 45 subjects will be enrolled at investigational sites in the United States (US) and China, though other countries may be added in the future. Approximately 45 subjects who meet the study entry criteria will randomly be assigned in a 1:1:1 ratio to receive 1 of 3 treatments: sirolimus 0.2% ointment, sirolimus 0.4% ointment, or placebo ointment. The randomization is stratified by site. Subjects, or a parent/guardian, will apply the study medication topically to the cutaneous angiofibromas on the face once daily at night before going to bed for 12 weeks. Subjects who complete the double-blind phase of the study, with an overall compliance rate >80% as determined by the dosing diary, will be offered entry into an open-label period for an additional 12 weeks.

The maximum study duration for each subject will be approximately 30 weeks and includes a screening period of up to 4 weeks, a blinded treatment period of 12 weeks, optional open-label period of 12 weeks, and a follow-up period of 2 weeks.

An interim analysis will be performed when all subjects have completed the double-blind phase (Visit 5 - Week 12). The data will be unblinded to assess for efficacy and results reported.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy males or non-pregnant females aged 2 to 21 years, inclusive, at the time of screening.
2. Diagnosis of TSC with visible facial angiofibromas of at least grade 3 up to grade 5, inclusive, based on the IGA.
3. Subjects with 3 or more isolated, measurable lesions of facial angiofibroma, with color grading score ≥2 for each of the 3 lesions.
4. Females of childbearing potential must have a negative urine pregnancy test (or a negative serum pregnancy test if a urine pregnancy test cannot be obtained) (For China, different pregnancy test would be followed) and if sexually active or become sexually active during the study, must agree to use an effective form of birth control for the duration of the study. Females using oral contraceptives must also use a barrier method of contraception during the study. Sexually active male subjects and/or their female partners should also use appropriate contraception.

   Effective contraception is defined as follows:
   * Oral/implant/injectable/transdermal/estrogenic vaginal ring contraceptives, intrauterine device, condom with spermicide, diaphragm with spermicide.
   * Abstinence or partner's vasectomy are acceptable if the female agrees to implement one of the other acceptable methods of birth control if her partner changes.
5. The subject and/or their parent or guardian must be willing and able to provide written informed consent/assent.
6. Willing and able to comply with all trial requirements.
7. Subject or parent/guardian must be able to complete the subject self-assessment survey and subject diary in English or another language into which the documents have been officially translated.
8. Subjects should be in good general health based on the subject's medical history, physical exam, and impression of the study doctor.

   Exclusion Criteria:
9. Has any chronic or acute medical condition, that in the opinion of the investigator, may pose a risk to the safety of the subject during the trial period, or may interfere with the assessment of safety or efficacy in this trial.
10. Has received oral therapy or topical therapy of an mTOR inhibitor (sirolimus, temsirolimus, or everolimus) within 1 month of Baseline or other dermatological treatment to facial angiofibromas within 1 month of baseline. (Sunscreen is expected to be used in this patient population and is not considered treatment.)
11. Is currently receiving any form of immunosuppression therapy or has previously experienced significant immune dysfunction.
12. Has a history of sensitivity to any component of the investigational product.
13. Is pregnant, plans to become pregnant during the course of the study, or is breastfeeding.
14. Has other dermatologic conditions, pigmentation, scarring, pigmented lesions or sunburn in the treatment area that would preclude or prevent adequate assessment of changes to their facial angiofibromas.
15. Has facial hair (e.g., beard, sideburns, mustache) that could interfere with study assessments.
16. Has had laser surgery or cryotherapy to facial angiofibromas within 6 months preceding study entry.
17. Requires the use of any concomitant medication that, in the investigator's opinion, has the potential to cause an adverse effect when given with the investigational product or will interfere with the interpretation of the study results (see Section 16.1 Appendix 1 for Potential Drug Interactions).
18. Has participated in another clinical trial or received an investigational product within 3 months prior to screening.

Ages: 2 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shoufeng Li, Ph.D, Study Director — Aucta Pharmaceuticals, Inc
Locations (8):
- United States (7):
  - Translational Genomics Research, Phoenix, Arizona
  - Children's Hospital of Los Angeles, Division of Neurology, Los Angeles, California
  - Children's Clinical Research Organization, Children's Hospital Colorado, Aurora, Colorado
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - LeBonheur Children's Hospital, Memphis, Tennessee
- Children's Hospital of Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Koenig MK, Hebert AA, Roberson J, Samuels J, Slopis J, Woerner A, Northrup H. Topical rapamycin therapy to alleviate the cutaneous manifestations of tuberous sclerosis complex: a double-blind, randomized, controlled trial to evaluate the safety and efficacy of topically applied rapamycin. Drugs R D. 2012 Sep 1;12(3):121-6. doi: 10.2165/11634580-000000000-00000. PMID 22934754
- [Background] Wheless JW, Almoazen H. A novel topical rapamycin cream for the treatment of facial angiofibromas in tuberous sclerosis complex. J Child Neurol. 2013 Jul;28(7):933-6. doi: 10.1177/0883073813488664. Epub 2013 May 16. PMID 23680945
- [Background] Wataya-Kaneda M, Tanaka M, Nakamura A, Matsumoto S, Katayama I. A topical combination of rapamycin and tacrolimus for the treatment of angiofibroma due to tuberous sclerosis complex (TSC): a pilot study of nine Japanese patients with TSC of different disease severity. Br J Dermatol. 2011 Oct;165(4):912-6. doi: 10.1111/j.1365-2133.2011.10471.x. PMID 21692771
- [Background] Tanaka M, Wataya-Kaneda M, Nakamura A, Matsumoto S, Katayama I. First left-right comparative study of topical rapamycin vs. vehicle for facial angiofibromas in patients with tuberous sclerosis complex. Br J Dermatol. 2013 Dec;169(6):1314-8. doi: 10.1111/bjd.12567. PMID 23909960
- [Background] Rapamune (sirolimus) complete prescribing information. Wyeth Pharmaceuticals Inc. October 2009

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were enrolled at 3-5 investigational sites in the United States.
Pre-assignment Details: At the time of study closure, a total of 28 participants were screened and 24 were randomized and received treatment. This study was early terminated due to another company receiving exclusivity.
Groups:
- Sirolimus 0.2%: Sirolimus 0.2% ointment applied topically once daily at bedtime for 12 weeks
- Sirolimus 0.4%: Sirolimus 0.4% ointment applied topically once daily at bedtime for 12 weeks
- Placebo: Placebo ointment applied topically once daily at bedtime for 12 weeks
Period: Double-Blind Phase
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Started | 7 | 8 | 9
Completed | 7 | 8 | 9
Not Completed | 0 | 0 | 0
Period: Open-label Phase
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Started | 7 | 8 | 9
Completed | 6 | 6 | 7
Not Completed | 1 | 2 | 2

BASELINE CHARACTERISTICS:
Population: [Not Specified]
Groups:
- Arm 1: Sirolimus 0.2% ointment applied topically once daily at bedtime for 12 weeks
- Arm 2: Sirolimus 0.4% ointment applied topically once daily at bedtime for 12 weeks
- Arm 3: Placebo ointment applied topically once daily at bedtime for 12 weeks
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 7 | 8 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.1 (2.73) | 13.1 (4.67) | 10.9 (3.44) | 12.0 (3.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 17
  Male | 3 | 2 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 2 | 5
  Not Hispanic or Latino | 6 | 6 | 7 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 2 | 3 | 2 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 5 | 5 | 6 | 16
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1
Height (cm) [Mean (Standard Deviation); unit: cm] | 154.8 (11.65) | 144.9 (23.04) | 141.2 (16.39) | 146.6 (18.02)
Weight (kg) [Mean (Standard Deviation); unit: kg] | 50.3 (20.08) | 41.3 (18.20) | 37.0 (9.37) | 42.3 (16.35)
BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 20.6 (6.52) | 18.7 (3.92) | 18.7 (2.85) | 19.2 (4.46)

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Participants Achieved at Least 2-grade Improvement
Description: The Investigator's Global Assessment (IGA) was recorded on a 5-point scale, 0 (minimum) to 5 (maximum) [0 = Clear skin with no signs of erythema and no disease related lesions, 1 = Slight redness with few disease related lesions, 2 = Greater than Grade 1; definite redness with scattered, some disease related lesions, 3 = Greater than Grade 2; marked redness, concentrated, many disease related lesions, 4 = Greater than Grade 3; very bright redness, confluent, highly concentrated disease related lesions, 5= Greater than Grade 4; fiery redness, very extensive disease related lesions covering very large area of the face]. A higher score indicates a more severe, worse outcome.
Time Frame: Double-blind phase and Open-label phase Weeks 4 and 12
Population: In the double-blind phase all randomized participants received study treatment and completed week 12 Investigator Global Assessment (IGA). In open-label phase, total of 19 participants completed week 24 (Open-label week 12) Investigator Global Assessment (IGA).
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  Primary Endpoint (>=2 point improvement) Week 12: No (N) | 6 | 6 | 9
  Primary Endpoint (>=2 point improvement) Week 12: Yes (Y) | 1 | 2 | 0
  Primary Endpoint (>=2 point improvement) Week 4: No (N) | 6 | 8 | 9
  Primary Endpoint (>=2 point improvement) Week 4: Yes (Y) | 1 | 0 | 0
  Primary Endpoint (>/=2 point improvement) (Open-label Week 4): number analyzed (Participants) | 7 | 6 | 9
  Primary Endpoint (>/=2 point improvement) (Open-label Week 4): No (N) | 6 | 5 | 7
  Primary Endpoint (>/=2 point improvement) (Open-label Week 4): Yes (Y) | 1 | 1 | 2
  Primary Endpoint (>=2 point improvement) (Open-label Week 12): number analyzed (Participants) | 6 | 6 | 7
  Primary Endpoint (>=2 point improvement) (Open-label Week 12): No (N) | 4 | 5 | 3
  Primary Endpoint (>=2 point improvement) (Open-label Week 12): Yes (Y) | 2 | 1 | 4

2. Primary Outcome: The Change in Baseline in Investigator's Global Assessment (IGA) by Visit
Description: The Investigator's Global Assessment (IGA) was recorded on a 5-point scale, 0 (minimum) to 5 (maximum) [0 = Clear skin with no signs of erythema and no disease related lesions, 1 = Slight redness with few disease related lesions, 2 = Greater than Grade 1; definite redness with scattered, some disease related lesions, 3 = Greater than Grade 2; marked redness, concentrated, many disease related lesions, 4 = Greater than Grade 3; very bright redness, confluent, highly concentrated disease related lesions, 5= Greater than Grade 4; fiery redness, very extensive disease related lesions covering very large area of the face]. A higher score indicates a more severe, worse outcome.
  Negative values indicate improvement (0 = no change, -1 = 1-point improvement, -2 = 2-point improvement)
Time Frame: Double-blind phase and Open-label phase Weeks 4 and 12
Population: In the double-blind phase, all randomized participants received study treatment and completed week 12 Investigator Global Assessment (IGA). In open-label phase, total of 19 participants completed week 24 (Open-label week 12) Investigator Global Assessment (IGA).
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  Change from Baseline in IGA by Visit: Week 4: 0 = No change from baseline | 2 | 4 | 8
  Change from Baseline in IGA by Visit: Week 4: -1 = 1- point improvement from baseline | 4 | 4 | 1
  Change from Baseline in IGA by Visit: Week 4: -2 = 2-point improvement from baseline | 1 | 0 | 0
  Change from Baseline in IGA by Visit: Week 4: -3 = 3-point improvement from baseline | 0 | 0 | 0
  Change from Baseline in IGA by Visit: Week 12: 0 = No change from baseline | 1 | 3 | 8
  Change from Baseline in IGA by Visit: Week 12: -1 = 1- point improvement from baseline | 5 | 3 | 1
  Change from Baseline in IGA by Visit: Week 12: -2 = 2-point improvement from baseline | 1 | 2 | 0
  Change from Baseline in IGA by Visit: Week 12: -3 = 3-point improvement from baseline | 0 | 0 | 0
  Change from Baseline in IGA by Visit: Open-label week 4: number analyzed (Participants) | 7 | 6 | 9
  Change from Baseline in IGA by Visit: Open-label week 4: 0 = No change from baseline | 1 | 2 | 1
  Change from Baseline in IGA by Visit: Open-label week 4: -1 = 1- point improvement from baseline | 5 | 3 | 6
  Change from Baseline in IGA by Visit: Open-label week 4: -2 = 2-point improvement from baseline | 1 | 1 | 2
  Change from Baseline in IGA by Visit: Open-label week 4: -3 = 3-point improvement from baseline | 0 | 0 | 0
  Change from Baseline in IGA by visit: Open-label week 12: number analyzed (Participants) | 6 | 6 | 7
  Change from Baseline in IGA by visit: Open-label week 12: 0 = No change from baseline | 0 | 2 | 0
  Change from Baseline in IGA by visit: Open-label week 12: -1 = 1- point improvement from baseline | 4 | 3 | 3
  Change from Baseline in IGA by visit: Open-label week 12: -2 = 2-point improvement from baseline | 1 | 1 | 3
  Change from Baseline in IGA by visit: Open-label week 12: -3 = 3-point improvement from baseline | 1 | 0 | 1

3. Secondary Outcome: The Percentage of Subjects With at Least 30% Improvement in the Facial Angiofibromas Severity Index (FASI) Score.
Description: The Facial Angiofibromas Severity Index (FASI) is derived from the measurements of erythema, average size, and lesion extension. The FASI score is the sum of scores of Erythema, Size, and Extension. Erythema was recorded on a 4-point grade scale from 0 (minimum) to 4 (maximum) [0 = clear skin with no signs of erythema, 1 = almost clear; slight redness, 3= moderate erythema; marked redness, 4= severe erythema; very bright redness]. Size was recorded on a 4-point grade scale from 0 (minimum) to 4 (maximum) [0 = no lesions, 1= few lesions, average size </= 2mm, 2 = scattered, some lesions, average lesion size >2-to </= 5 mm, 3 = concentrated, many lesions, average lesion size > 5mmg to </= 10mm, 4 = confluent, highly concentrated lesions]. Extension was recorded on a grade scale of 0 (minimum), 2, and 3 (maximum) [0 = no lesions, 2 = </= 50% of the cheek surface, 3 = >50% of the cheek surface]. A higher score for Erythema, Size, and Extension means a more severe, worse outcome.
Time Frame: Double-blind phase Weeks 4 and 12 and Open-label phase Week 12
Population: [Not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  >=30% Improvement in FASI Score Week 4: No (N) | 5 | 6 | 9
  >=30% Improvement in FASI Score Week 4: Yes (Y) | 2 | 2 | 0
  >=30% Improvement in FASI Score Week 12: No (N) | 5 | 5 | 9
  >=30% Improvement in FASI Score Week 12: Yes (Y) | 2 | 3 | 0
  >= 30% Improvement in FASI Score: Open-label week 12: number analyzed (Participants) | 5 | 6 | 6
  >= 30% Improvement in FASI Score: Open-label week 12: No (N) | 3 | 5 | 3
  >= 30% Improvement in FASI Score: Open-label week 12: Yes (Y) | 2 | 1 | 3

4. Secondary Outcome: Facial Angifibromas Severity Index (FASI) Score
Description: as for outcome 3
Time Frame: Baseline, Double blind phase weeks 4 and 12 and Open-label week 12
Population: [Not specified]
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
score on a scale
  Baseline FASI Total Score | 6.86 (1.35) | 7.38 (1.19) | 7.89 (1.27)
  Week 4 FASI Total Score | 5.71 (1.25) | 6.5 (1.69) | 7.33 (1.32)
  Week 12 FASI Total Score | 5.57 (0.98) | 5.75 (1.39) | 7 (1.58)
  Open-label week 12 FASI Total Score: number analyzed (Participants) | 5 | 5 | 6
  Open-label week 12 FASI Total Score | 5 (1) | 6 (0.63) | 5.33 (1.51)

5. Secondary Outcome: The Percentage of Subjects Achieved at Least 2-grade Improvement in Categorical Lesion Counts by Visit
Description: Lesion counts are measured based on categories 0 to 4 [0 = no lesion, 1 = <25 lesions, 2 = 25 to 50 lesions, 3 = 51 to 75 lesions, 4 = > 75 lesions]
Time Frame: Double blind phase Weeks 4 and 12 and Open-label phase Week 12
Population: [Not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  >=2 grade improvement in lesion: Week 4: No (N) | 6 | 7 | 9
  >=2 grade improvement in lesion: Week 4: Yes (N) | 1 | 1 | 0
  >=2 grade improvement in lesion: Week 12: No (N) | 6 | 7 | 9
  >=2 grade improvement in lesion: Week 12: Yes (N) | 1 | 1 | 0
  >=2 grade improvement in lesion: Open-label week 12: number analyzed (Participants) | 5 | 6 | 6
  >=2 grade improvement in lesion: Open-label week 12: No (N) | 4 | 5 | 4
  >=2 grade improvement in lesion: Open-label week 12: Yes (N) | 1 | 1 | 2

6. Secondary Outcome: Change From Baseline in Lesion Counts
Description: Lesion counts are measured based on categories 0 to 4 (0 = no lesion, 1 = <25 lesions, 2 = 25 to 50 lesions, 3 = 51 to 75 lesions, 4 = > 75 lesions) Negative values indicate improvement (0 = no change, -1 = 1-point improvement, -2 = 2-point improvement)
Time Frame: Double blind phase weeks 4 and 12 and open-label phase week 12
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  Change from Baseline in lesion counts by visit: Week 4: 0 = No change from baseline | 6 | 5 | 8
  Change from Baseline in lesion counts by visit: Week 4: -1 = 1-point improvement from baseline | 0 | 2 | 1
  Change from Baseline in lesion counts by visit: Week 4: -2 = 2-point improvement from baseline | 1 | 1 | 0
  Change from Baseline in lesion counts by visit: Week 4: -3 = 3-point improvement from baseline | 0 | 0 | 0
  Change from Baseline in lesion counts by visit: Week 12: 0 = No change from baseline | 3 | 5 | 9
  Change from Baseline in lesion counts by visit: Week 12: -1 = 1-point improvement from baseline | 3 | 2 | 0
  Change from Baseline in lesion counts by visit: Week 12: -2 = 2-point improvement from baseline | 1 | 0 | 0
  Change from Baseline in lesion counts by visit: Week 12: -3 = 3-point improvement from baseline | 0 | 1 | 0
  Change from baseline in lesion counts by visit: Open-label week 12: number analyzed (Participants) | 5 | 6 | 6
  Change from baseline in lesion counts by visit: Open-label week 12: 0 = No change from baseline | 2 | 2 | 2
  Change from baseline in lesion counts by visit: Open-label week 12: -1 = 1-point improvement from baseline | 2 | 3 | 2
  Change from baseline in lesion counts by visit: Open-label week 12: -2 = 2-point improvement from baseline | 1 | 0 | 2
  Change from baseline in lesion counts by visit: Open-label week 12: -3 = 3-point improvement from baseline | 0 | 1 | 0

7. Secondary Outcome: The Percentage of Subjects Achieved at Least 2-grade Improvement in Lesion Elevation.
Description: The degree of lesion elevation is assessed on categories 0 to 4 (0 = no elevation over normal skin, 1 = possible but difficult to ascertain whether there is slight elevation above normal skin, 2 = slight but definite elevation, 3 = moderate elevation, 4 = marked elevation).
Time Frame: Double blind phase weeks 4 and 12 and open-label phase week 12
Population: [Not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  >=2 grade improvement in lesion elevation: Week 4: No (N) | 6 | 8 | 9
  >=2 grade improvement in lesion elevation: Week 4: Yes (Y) | 1 | 0 | 0
  >=2 grade improvement in lesion elevation: Week 12: No (N) | 6 | 8 | 9
  >=2 grade improvement in lesion elevation: Week 12: Yes (Y) | 1 | 0 | 0
  >=2 grade improvement in lesion elevation: Open-label week 12: number analyzed (Participants) | 5 | 6 | 6
  >=2 grade improvement in lesion elevation: Open-label week 12: No (N) | 4 | 5 | 6
  >=2 grade improvement in lesion elevation: Open-label week 12: Yes (Y) | 1 | 1 | 0

8. Secondary Outcome: The Change From Baseline in Lesion Elevation
Description: The degree of lesion elevation is assessed on categories 0 to 4 (0 = no elevation over normal skin, 1 = possible but difficult to ascertain whether there is slight elevation above normal skin, 2 = slight but definite elevation, 3 = moderate elevation, 4 = marked elevation) Negative values indicate improvement (0 = no change, -1 = 1-point improvement, -2 = 2-point improvement) One participant with baseline elevation grade of 1 improved to grade 0 at week 4. This participant is counted as improvement in lesion elevation. This participant was back to grade 1 at week 12 and open-label week 12.
Time Frame: Double blind phase weeks 4 and 12 and open-label phase week 12
Population: [Not Specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  Change from Baseline in lesion elevation: Week 4: 0 = No change from baseline | 4 | 4 | 8
  Change from Baseline in lesion elevation: Week 4: -1 = 1-point improvement from baseline | 2 | 4 | 1
  Change from Baseline in lesion elevation: Week 4: -2 = 2-point improvement from baseline | 1 | 0 | 0
  Change from Baseline in lesion elevation: Week 12: 0 = No change from baseline | 3 | 4 | 9
  Change from Baseline in lesion elevation: Week 12: -1 = 1-point improvement from baseline | 3 | 4 | 0
  Change from Baseline in lesion elevation: Week 12: -2 = 2-point improvement from baseline | 1 | 0 | 0
  Change from baseline in lesion elevation: Open-label week 12: number analyzed (Participants) | 5 | 6 | 6
  Change from baseline in lesion elevation: Open-label week 12: 0 = No change from baseline | 2 | 3 | 3
  Change from baseline in lesion elevation: Open-label week 12: -1 = 1-point improvement from baseline | 2 | 2 | 3
  Change from baseline in lesion elevation: Open-label week 12: -2 = 2-point improvement from baseline | 1 | 1 | 0

9. Secondary Outcome: The Percentage of Subjects Achieved at Least 2-grade Improvement in the Subject Self-assessment Survey
Description: Subject self- assessment survey was based on categories 0 to 4 (0 = no redness and no disease related lesions, 1 = very mild redness with few very small bumps, 2 = mild redness with many small and medium sized bumps, 3 = moderate redness with many small and medium sized bumps, 4 = severe redness with numerous small, medium, and large sized bumps)
Time Frame: Double blind phase weeks 4 and 12 and open-label phase weeks 4 and 12
Population: [Not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  >=2 grade improvement in self-assessment: Week 4: No (N) | 6 | 7 | 9
  >=2 grade improvement in self-assessment: Week 4: Yes (Y) | 1 | 1 | 0
  >=2 grade improvement in self-assessment: Week 12: No (N) | 5 | 6 | 8
  >=2 grade improvement in self-assessment: Week 12: Yes (Y) | 2 | 2 | 1
  >=2 grade improvement in self-assessment: open-label week 4: number analyzed (Participants) | 7 | 6 | 9
  >=2 grade improvement in self-assessment: open-label week 4: No (N) | 5 | 2 | 8
  >=2 grade improvement in self-assessment: open-label week 4: Yes (Y) | 2 | 4 | 1
  >=2 grade improvement in self-assessment: open-label week 12: number analyzed (Participants) | 6 | 6 | 7
  >=2 grade improvement in self-assessment: open-label week 12: No (N) | 3 | 3 | 4
  >=2 grade improvement in self-assessment: open-label week 12: Yes (Y) | 3 | 3 | 3

10. Secondary Outcome: Change From Baseline in Self-Assessment
Description: Subject self- assessment survey was based on categories 0 to 4 (0 = no redness and no disease related lesions, 1 = very mild redness with few very small bumps, 2 = mild redness with many small and medium sized bumps, 3 = moderate redness with many small and medium sized bumps, 4 = severe redness with numerous small, medium, and large sized bumps) Negative values indicate improvement (0 = no change, -1 = 1-point improvement, -2 = 2-point improvement)
Time Frame: Double blind phase weeks 4 and 12 and open label phase weeks 4 and 12
Population: [Not specified]
Measure: Count of Participants; unit: Participants
Arm/Group | Sirolimus 0.2% | Sirolimus 0.4% | Placebo
Number analyzed (Participants) | 7 | 8 | 9
Participants
  Change from baseline in self-assessment: Week 4: 1 = 1-point worsening from baseline | 0 | 0 | 0
  Change from baseline in self-assessment: Week 4: 0 = No change from baseline | 3 | 3 | 8
  Change from baseline in self-assessment: Week 4: -1 = 1-point improvement from baseline | 3 | 4 | 1
  Change from baseline in self-assessment: Week 4: -2 = 2-point improvement from baseline | 1 | 1 | 0
  Change from baseline in self-assessment: Week 4: -3 = 3-point improvement from baseline | 0 | 0 | 0
  Change from Baseline in self-assessment: Week 12: 1 = 1-point worsening from baseline | 0 | 0 | 0
  Change from Baseline in self-assessment: Week 12: 0 = No change from baseline | 1 | 1 | 6
  Change from Baseline in self-assessment: Week 12: -1 = 1-point improvement from baseline | 4 | 5 | 2
  Change from Baseline in self-assessment: Week 12: -2 = 2-point improvement from baseline | 1 | 2 | 1
  Change from Baseline in self-assessment: Week 12: -3 = 3-point improvement from baseline | 1 | 0 | 0
  Change from baseline in self- assessment: open-label week 14: number analyzed (Participants) | 7 | 6 | 9
  Change from baseline in self- assessment: open-label week 14: 1 = 1-point worsening from baseline | 0 | 0 | 0
  Change from baseline in self- assessment: open-label week 14: 0 = No change from baseline | 1 | 2 | 3
  Change from baseline in self- assessment: open-label week 14: -1 = 1-point improvement from baseline | 4 | 0 | 5
  Change from baseline in self- assessment: open-label week 14: -2 = 2-point improvement from baseline | 2 | 3 | 1
  Change from baseline in self- assessment: open-label week 14: -3 = 3-point improvement from baseline | 0 | 1 | 0
  Change from baseline in self-assessment: open-label week 12: number analyzed (Participants) | 6 | 6 | 7
  Change from baseline in self-assessment: open-label week 12: 1 = 1-point worsening from baseline | 0 | 0 | 1
  Change from baseline in self-assessment: open-label week 12: 0 = No change from baseline | 0 | 1 | 1
  Change from baseline in self-assessment: open-label week 12: -1 = 1-point improvement from baseline | 3 | 2 | 2
  Change from baseline in self-assessment: open-label week 12: -2 = 2-point improvement from baseline | 2 | 3 | 3
  Change from baseline in self-assessment: open-label week 12: -3 = 3-point improvement from baseline | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 weeks
Groups:
- Double-Blind: Sirolimus 0.2%; Open-label: Sirolimus 0.2%: Sirolimus 0.2% ointment applied topically once daily at bedtime for 12 weeks
- Double-Blind: Sirolimus 0.4%; Open-label: Sirolimus 0.4%: Sirolimus 0.4% ointment applied topically once daily at bedtime for 12 weeks
- Double-Blind: Placebo; Open-label: Placebo: Placebo ointment applied topically once daily at bedtime for 12 weeks
Arm/Group | Double-Blind: Sirolimus 0.2% | Double-Blind: Sirolimus 0.4% | Double-Blind: Placebo | Open-label: Sirolimus 0.2% | Open-label: Sirolimus 0.4% | Open-label: Placebo
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/8 | 0/9 | 0/7 | 0/7 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/8 | 1/9 | 1/7 | 1/7 | 0/9
Other Adverse Events (participants affected / at risk) | 6/7 | 5/8 | 4/9 | 1/7 | 5/7 | 4/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind: Sirolimus 0.2% (N=7) | Double-Blind: Sirolimus 0.4% (N=8) | Double-Blind: Placebo (N=9) | Open-label: Sirolimus 0.2% (N=7) | Open-label: Sirolimus 0.4% (N=7) | Open-label: Placebo (N=9)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Treatment-emergent Serious Adverse Event
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Treatment-emergent Serious Adverse Event
Psychotic disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Treatment-emergent Serious Adverse Event
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double-Blind: Sirolimus 0.2% (N=7) | Double-Blind: Sirolimus 0.4% (N=8) | Double-Blind: Placebo (N=9) | Open-label: Sirolimus 0.2% (N=7) | Open-label: Sirolimus 0.4% (N=7) | Open-label: Placebo (N=9)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application site reaction (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Obsessive thoughts (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dsymenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT03363763/Prot_SAP_000.pdf